CLINICAL TRIAL: NCT00060580
Title: Measurement of Macular Pigment With Resonant Raman Backscattering Spectroscopy
Brief Title: Raman Scattering Spectroscopy to Measure Macular Pigment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030156; 03-EI-0156
Record Dates: First submitted 2003-05-07; First posted 2003-05-08 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-03

CONDITIONS: Raman Spectroscopy
Keywords: Retinal Measurements; Lutein in Vivo; Raman Spectroscopy; Retinal Measurements of Lutein in Vivo in the Human Eye; Healthy Volunteer; HV
MeSH Terms: interventions — Spectrum Analysis, Raman

INTERVENTIONS:
Procedure: Raman scattering spectroscopy

SUMMARY:
This study will evaluate the ease and reliability of Raman scattering spectroscopy, a new technique to measure the amount of the pigment lutein in the retina, the light-sensitive tissue lining the back of the eye. The highest concentrations of lutein are in the center of the retina, called the macula, which is the area most important for fine, detailed vision. The functions of lutein are not fully known. Besides absorbing blue light, it may help protect against abnormal changes in the retina, such as age-related macular degeneration. Until recently, lutein was measured using long, cumbersome, and difficult tests. This study will evaluate a new instrument that provides faster measurements. It will be tested under different conditions, such as wearing or not wearing glasses or contact lenses, or dilating or not dilating the pupil of the eye.

Healthy normal volunteers between 20 and 65 years of age may be eligible for this study, which involves two visits to the NIH Clinical Center, as follows:

Visit 1 - Screening

* Medical history and physical examination, including measurement of vital signs (blood pressure, pulse, temperature, and breathing rate), and examination of the head and neck, heart and lungs, and arms and legs.
* Eye examination, including eye chart test, eye pressure measurement, examination of pupils and eye movements, and examination of the retina (back part of the eye) using a strong light and magnifying lens after dilation of the pupils.
* Raman scattering spectroscopy to measure lutein. For this test, the subject looks with one eye at a brief, bright flash of bluish light (similar to a flashbulb light) from a laser. This is repeated several times. Subjects who wear glasses or contact lenses for distance vision will be tested without them and then again with a lens in front of the eye. Subjects who do not wear glasses or contact lenses will be tested before and after dilation of the pupil.
* Contrast sensitivity to assess ability to identify an object from the background and to see everyday objects. The subject looks at and identifies a variety of objects of different shapes and sizes.
* Color vision to determine the ability to identify different shades of color. The subject arranges a line of colorful discs, similar to checkers, in order of similar shades.

Visit 2 - Repeat Spectroscopy

Subjects return 1 week after the screening visit for a repeat Raman scattering spectroscopy to evaluate the precision of the measurements.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the degree of variability in retinal measurements of lutein, a carotenoid macular pigment of human retina in normal volunteers, with a new and novel technique of resonant Raman scattering spectroscopy. This technique is generally more objective than psychophysical techniques used for lutein measurements, such as heterochromatic flicker photometry. Raman scattering spectroscopy is non-invasive and the levels of ocular exposure to argon laser light used in this technique are well below the safety limits recommended by the American National Standards Institute.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Men and women between 18 and 75 years of age.
2. Corrected visual acuity of 20/30 or better.
3. Ability to understand and sign an informed consent form prior to enrollment.

EXCLUSION CRITERIA:

1. Ocular disease, including significant explained or unexplained visual field loss.
2. Ocular media opacities.
3. History of epilepsy or light-triggered convulsions.
4. A maximal pupillary dilation of less than 7 mm.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-05; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bone RA, Landrum JT, Tarsis SL. Preliminary identification of the human macular pigment. Vision Res. 1985;25(11):1531-5. doi: 10.1016/0042-6989(85)90123-3. PMID 3832576
- [Background] Landrum JT, Bone RA, Joa H, Kilburn MD, Moore LL, Sprague KE. A one year study of the macular pigment: the effect of 140 days of a lutein supplement. Exp Eye Res. 1997 Jul;65(1):57-62. doi: 10.1006/exer.1997.0309. PMID 9237865
- [Background] Seddon JM, Ajani UA, Sperduto RD, Hiller R, Blair N, Burton TC, Farber MD, Gragoudas ES, Haller J, Miller DT, et al. Dietary carotenoids, vitamins A, C, and E, and advanced age-related macular degeneration. Eye Disease Case-Control Study Group. JAMA. 1994 Nov 9;272(18):1413-20. PMID 7933422